CLINICAL TRIAL: NCT03059615
Title: A Phase 2a, Open-Label, Two Stage Study: Stage A: Dose-Range Finder Study to Assess the Safety and Efficacy of Two Doses of Nerofe and Two Doses of Nerofe in Combination With Doxorubicin in Subjects With Acute Myelogenous Leukemia or High Risk Myelodysplastic Syndrome (AML/High Risk MDS). Stage B: Dose Confirmation Study to Assess the Safety and Efficacy of Nerofe or Nerofe in Combination With Doxorubicin in Subjects With AML/ High Risk MDS
Brief Title: A Phase 2a, Open-Label, Two Stage Study of Nerofe or Nerofe With Doxorubicin in Subjects With AML or MDS
Status: Withdrawn | Phase: Phase 2 | Type: Interventional
Why Stopped: No recruitment since initiation
Sponsor: Immune System Key Ltd (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: ISK-N102
Record Dates: First submitted 2017-02-09; First posted 2017-02-23 (Actual); Last update posted 2020-07-31 (Actual); Status verified 2020-07

CONDITIONS: Acute Myelogenous Leukemia; Myelodysplastic Syndromes
MeSH Terms: conditions — Leukemia, Myeloid, Acute; Myelodysplastic Syndromes | interventions — tumor-cells apoptosis factor, human; Doxorubicin

STUDY DESIGN:
Intervention Model Description: 2 stage study:
  1. Dose Range Finder (4 treatment arms)
  2. Dose Confirmation (1 chosen treatment arm)
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- Nerofe 48mg/m2 (Experimental): 48mg/m2 IV Nerofe - three times a week
  Interventions: Drug: Nerofe
- Nerofe 96mg/m2 (Experimental): 96mg/m2 IV Nerofe - three times a week
  Interventions: Drug: Nerofe
- Nerofe 48mg/m2 + Doxorubicin 10mg/m2 (Experimental): 48mg/m2 IV Nerofe + Doxorubicin 10mg/m2 - once a week
  Interventions: Drug: Nerofe; Drug: Doxorubicin
- Nerofe 96mg/m2 + Doxorubicin 10mg/m2 (Experimental): 96mg/m2 IV Nerofe + Doxorubicin 10mg/m2 - once a week
  Interventions: Drug: Nerofe; Drug: Doxorubicin

INTERVENTIONS:
Drug: Nerofe — Nerofe is a first-in-class hormone-peptide with cancer suppressive properties. Nerofe is a derivative of the human hormone-peptide Tumor-Cells Apoptosis Factor (TCApF). It contains 14 amino-acids. Binding Nerofe to the T1/ST2 receptor caused a rapid activation both of Caspase 8 and Bcl-2 mediated downstream in proliferating cancer cells.
Drug: Doxorubicin — Doxorubicin is an anthracycline antibiotic with antineoplastic activity. Doxorubicin, isolated from the bacterium Streptomyces peucetius var. caesius, is the hydroxylated congener of daunorubicin. Doxorubicin intercalates between base pairs in the DNA helix, thereby preventing DNA replication and ultimately inhibiting protein synthesis.
  Arms: Nerofe 48mg/m2 + Doxorubicin 10mg/m2; Nerofe 96mg/m2 + Doxorubicin 10mg/m2

SUMMARY:
This is a Phase 2a, Open-label, one arm study in which the eligible patients will be treated with IV Nerofe, three times a week in 28 days cycles (up to 12 cycles).

Evaluation will include safety procedures, blood level of study drug in certain time points, immune system response and tests checking the mechanism of the drug action.

DETAILED DESCRIPTION:
Nerofe is a first-in-class hormone peptide with cancer suppressive properties. It works in three mechanisms of action. The purpose of this research is to study Nerofe's effect in patients diagnosed with AML and MDS.

ELIGIBILITY:
Inclusion Criteria

1. Males and females ≥18 years of age.
2. Either:

   * AML patients, who are not candidates for aggressive therapy and/or stem cell transplant (usually the elderly patients), or
   * Low and high prognostic risk MDS patients (according to the IPSS-R classification), resistant or relapsing following at least 1 course of hypo-methylation therapy.
3. Anti-tumor (in this case the anti-MDS or anti-leukemic) effect can be measured according to the IWG criteria (Appendices B, C).
4. Eastern Cooperative Oncology Group (ECOG) Performance Status of ≤ 2
5. Acceptable clinical laboratory values at screening, as indicated by:

   * Absolute neutrophil count ≥ 1,000/mm3;
   * Platelets ≥ 50,000/mm3;
   * Hemoglobin ≥ 6.5 g/dl ;
   * Total bilirubin ≤ 1.5 × the upper limit of normal (ULN);
   * AST (SGOT) ≤ 2.5 × the ULN;
   * ALT (SGPT) ≤ 2.5 × the ULN;
   * Serum creatinine ≤ 1.5 mg/dL or a measured creatinine clearance 60 mL/min and above
6. Negative serum β hCG test in women of childbearing potential
7. Women of childbearing potential must agree to use dual contraceptive methods while on study drug and for 3 months afterward.
8. Men who partner with a woman of childbearing potential must agree to use effective, dual contraceptive methods while on study drug and for 3 months afterward.
9. Willing and able to provide written acceptance that during the trial, bone marrow examination should be performed, with cytogenetics. Bone marrow examination will be performed at Screening, Cycle 3, every odd subsequent cycles and End of Dosing Visit (as per PI and Medical Monitor decision).
10. Bone marrow positive for ST2 receptor expression.
11. Willing and able to provide written Informed Consent and comply with the requirements of the study

Exclusion Criteria

1. Any chemotherapy, immunomodulatory drug therapy, anti-neoplastic hormonal therapy 30 days prior to study entry and , immunosuppressive therapy, prednisone > 20 mg/day, or any equivalent corticosteroids during the last six months.
2. Erythroid stimulating agents are allowed until one day prior to treatment initiation with study drug.
3. Presence of an acute toxicity of prior chemotherapy, with the exception of alopecia or peripheral neuropathy, that has not resolved to ≤ Grade 2, as determined by NCI CTCAE v 4.0
4. Receipt of >1 prior regimen of genotoxic therapy.
5. Previous bone marrow transplantation.
6. Life expectancy <12 weeks.
7. RBC transfusions for at least 1 week and platelet transfusions for at least 3 days prior to study entry.
8. Known human immunodeficiency virus (HIV) or acquired immunodeficiency syndrome-related illness (AIDS).
9. Known active hepatitis B or C or other active liver disease
10. Active infection requiring systemic therapy.
11. Unstable Insulin-dependent diabetes mellitus (IDDM), defined by one or more hospitalization (including ER visits) due to high or low blood glucose levels within the last 6 months.
12. History of any of the following within 12 months prior to initiation of study drug: Uncontrolled congestive heart failure (New York Heart Association Classification 3 or 4), unstable angina, myocardial infarction, cerebrovascular accident, coronary/peripheral artery bypass graft surgery, transient ischemic attack, or pulmonary embolism (within the last 6 month).
13. Uncontrolled hypertension and change in treatment regimen within the last month prior to screening.
14. Risk of syncope, in the judgment of the Principle Investigator, according to the patient's history of Syncope.
15. History of ongoing cardiac dysrhythmias requiring drug treatment.
16. Malignancies during the last yearexcept for skin non-melanomatous tumors and thyroid carcinomas..
17. Any known severe multiple allergy or acute allergic reaction.
18. Use of any investigational agents within 4 weeks or 5 half-lives of initiation of study drug.
19. Pregnant or lactating women.
20. Any severe, acute, or chronic medical or psychiatric condition, or laboratory abnormality that may increase the risk associated with study participation or study drug administration, may interfere with the informed consent process and/or with compliance with the requirements of the study, or may interfere with the interpretation of study results and, in the investigator's opinion, would make the patient inappropriate for entry into this study.

    For combination therapy only:
21. Impaired cardiac function defined as left ventricular ejection fraction (LVEF) ≤ 55 % as measured by ECHO.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2018-10-25 (Actual); Primary Completion 2020-07-26 (Actual); Study Completion 2020-07-26 (Actual)

PRIMARY OUTCOMES:
Assessing change in IWG Criteria to evaluate response to Nerofe treatment (with or without Doxorubicin) for AML subjects | At end of Cycles 2, 4, 6, 8, 10, 12 (Cycle length 28 Days)
  Bone Marrow samples and CBC will be done every 2 cycles
Assessing changes in R-IPSS (Revised International Prognostic Scoring System) Score to evaluate response to Nerofe treatment (with or without Doxorubicin) for MDS patients. A calculation of several variables. | At end of Cycles 2, 4, 6, 8, 10, 12 (Cycle length 28 Days)
  Bone Marrow samples to measure percentage of blasts (%). Range 0-30% (the higher the percentage the worse outcome).
Assessing changes in R-IPSS (Revised International Prognostic Scoring System) Score to evaluate response to Nerofe treatment (with or without Doxorubicin) for MDS patients. A calculation of several variables. | At end of Cycles 2, 4, 6, 8, 10, 12 (Cycle length 28 Days)
  Complete Blood Count (CBC) to measure hemoglobin (g/dL). Range 4-20 (4 worse outcome and 20 best outcome).
Assessing changes in R-IPSS (Revised International Prognostic Scoring System) Score to evaluate response to Nerofe treatment (with or without Doxorubicin) for MDS patients. A calculation of several variables. | At end of Cycles 2, 4, 6, 8, 10, 12 (Cycle length 28 Days)
  Complete Blood Count (CBC) to measure absolute neutrophil count (x10^9/L). Range 0-15 (the higher the score the better outcome).
Assessing changes in R-IPSS (Revised International Prognostic Scoring System) Score to evaluate response to Nerofe treatment (with or without Doxorubicin) for MDS patients. A calculation of several variables. | At end of Cycles 2, 4, 6, 8, 10, 12 (Cycle length 28 Days)
  Complete Blood Count (CBC) to measure platelets (x10^9/L). Range 0-2000 (the higher the score the better outcome)
Assessing changes in R-IPSS (Revised International Prognostic Scoring System) Score to evaluate response to Nerofe treatment (with or without Doxorubicin) for MDS patients. A calculation of several variables. | At end of Cycles 2, 4, 6, 8, 10, 12 (Cycle length 28 Days)
  Measuring cytogenetic abnormalities. Range from very good (0) to very poor (4)
Safety as determined by frequency, nature and severity of adverse events | 13 months
  Per CTCAE v4.0

SECONDARY OUTCOMES:
Pharmacokinetic behavior of Nerofe: Maximum Plasma Concentration (Cmax) | At cycles 1 and 2 (Cycle length 28 days)
  Done at Cycle 1 and 2: pre-dose, 15 minutes, 1, 2, 4, 6, 8 and 24 hours.
Pharmacokinetic behavior of Nerofe: Minimum Plasma Concentration (Cmin) | At cycles 1 and 2 (Cycle length 28 days)
  Done at Cycle 1 and 2: pre-dose, 15 minutes, 1, 2, 4, 6, 8 and 24 hours.
Pharmacokinetic behavior of Nerofe: Area Under the Curve (AUC) | At cycles 1 and 2 (Cycle length 28 days)
  Done at Cycle 1 and 2: pre-dose, 15 minutes, 1, 2, 4, 6, 8 and 24 hours.
Pharmacokinetic behavior of Nerofe: Tmax | At cycles 1 and 2 (Cycle length 28 days)
  Done at Cycle 1 and 2: pre-dose, 15 minutes, 1, 2, 4, 6, 8 and 24 hours.
Pharmacodynamic analysis of changes from baseline in levels of circulating cytokines | Every cycle (Cycle length 28 days)
  At Cycle 1 and 2 on Day 1 and Day 15 and on day 1 of each consecutive cycle (up to 12 cycles)
Pharmacodynamic analysis of changes from baseline in levels of soluble T1/ST2 receptor | Every cycle (Cycle length 28 days)
  At Cycle 1 and 2 on Day 1 and Day 15 and on day 1 of each consecutive cycle (up to 12 cycles)
Pharmacodynamic analysis of changes from baseline in PBMCs' T1/ST2 receptor expression | Every cycle (Cycle length 28 days)
  At Cycle 1 and 2 on Day 1 and Day 15 and on day 1 of each consecutive cycle (up to 12 cycles)

CONTACTS AND LOCATIONS:
Overall Officials: Yoram Devary, Study Director — Immune System Key Ltd
Locations (2):
- Israel (2):
  - Rabin Medical Center, Petah Tikva
  - Kaplan Medical Center, Rehovot

IPD SHARING:
Plan to Share IPD: No